CLINICAL TRIAL: NCT06947746
Title: A Single-arm Clinical Study Assessing the Safety, Tolerability, and Preliminary Efficacy of a Single Intra-Articular Injection of hiSCs for Rheumatoid Arthritis Treatment
Brief Title: HiSCs in the Treatment of Rheumatoid Arthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Xu huji, Professor and Chief Physician, Head of the Department of Rheumatology and Immunology, Shanghai Changzheng Hospital., Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HWHY-hiSC-01
Record Dates: First submitted 2025-03-26; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Sertoli cells; Rheumatoid Arthritis (RA); intra-articular injection; hiSCs
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- hiSCs treatment (Experimental): hiSCs，human induced Sertoli-like cells
  Interventions: Biological: hiSCs

INTERVENTIONS:
Biological: hiSCs — hiSCs are derived from human induced pluripotent stem cells and exhibit immunomodulatory properties.

SUMMARY:
This trial is a single-center, single-arm exploratory clinical study aimed at assessing the safety, tolerability, and preliminary efficacy of a single intra-articular injection of hiSCs for the treatment of rheumatoid arthritis.

DETAILED DESCRIPTION:
This trial is a single-center, single-arm exploratory clinical study aimed at assessing the safety, tolerability, and preliminary efficacy of a single intra-articular injection of hiSCs for the treatment of rheumatoid arthritis.

In this trial, participants who have given informed consent will be screened to determine their eligibility according to the inclusion and exclusion criteria. The study intervention consists of a single injection of hiSCs, and the primary endpoint will be assessed during the 24-week follow-up visit after the cell injection.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria

1. Voluntarily sign the informed consent;
2. Male or female aged 18-65 years (inclusive) at the time of signing the informed consent;
3. Diagnosis of RA for ≥3 months according to the ACR/EULAR 2010 Rheumatoid Arthritis Classification Criteria at the screening visit;
4. At the screening visit, presence of recurrent swelling and pain in at least one knee, with a WOMAC pain score ≥4, synovial inflammation confirmed by joint ultrasound, and no significant improvement following 3 months of anti-RA treatment (including prior use of MTX standard therapy, biologics, or small molecule targeted drugs);
5. Subjects must have received csDMARD therapy for ≥3 months, with a stable dose for ≥4 weeks prior to screening;
6. Background treatment with stable-dose MTX standard therapy, biologics, or small molecule targeted drugs, either alone or in combination, is permitted;
7. The following csDMARDs, either alone or in combination, are permitted as background treatment, provided the dose has been stable for ≥4 weeks prior to screening: oral or IV MTX (10-25 mg/week; for subjects intolerant to doses ≥10 mg/week, the dose should be ≥7.5 mg/week), SAS (≤3 g/day), hydroxychloroquine (≤400 mg/day), and LEF (≤20 mg/day);
8. Stable-dose NSAIDs are permitted, provided the dose has remained stable for ≥2 weeks prior to screening;
9. CRP or hsCRP levels exceeding the upper limit of normal at the screening visit;
10. All females of childbearing potential must have a negative blood pregnancy test within 7 days prior to treatment initiation and must not be breastfeeding. Females not of childbearing potential may be exempt from the pregnancy test and contraception if they meet one of the following criteria: age ≥50 years,not receiving hormone therapy, and at least 12 months of amenorrhea, or documented surgical sterilization. All enrolled patients (regardless of gender) must use at least one highly effective method of contraception, including adequate barrier methods, throughout the study duration;
11. Subjects must be in good overall health, able to ambulate independently (excluding those requiring a wheelchair, walker, or crutches);
12. Willingness and ability to adhere to scheduled visits, treatment regimens, laboratory tests, and other study-related procedures.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria will be excluded from this study：

1. Presence of other immune-mediated disorders at the baseline visit that may interfere with the administration or efficacy evaluation of the study intervention;
2. History or current evidence of clinically significant cardiovascular, neuropsychiatric, renal, hepatic, immune, or endocrine disorders (including uncontrolled diabetes or thyroid disease), abnormal laboratory findings, or conditions requiring medications prohibited by the study protocol. "Clinically significant" refers to conditions that, in the investigator's judgment, may jeopardize subject safety or impact efficacy or safety analyses if the disease/condition exacerbates during the study;
3. Subjects with positive test results for human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), or syphilis (refer to laboratory tests for details);
4. Evidence of active tuberculosis (TB) or a history of active TB without adequate documented treatment;
5. Any other acute or chronic disorder leading to coagulation dysfunction that, in the investigator's judgment, may compromise patient safety and/or interfere with the evaluation of target knee outcomes;
6. Clinically significant infection within 1 month prior to the screening visit (requiring hospitalization and parenteral administration of antibiotics, antivirals, antifungals, etc., for ≥3 days) or active infection being treated during the screening period;
7. Infection in the target knee within 3 months before baseline;
8. Intra-articular corticosteroid or other drug injections in the target knee within 3 months before baseline;
9. History of knee injury or prior knee surgery in the target knee within 1 year prior to the baseline visit;
10. Serum transaminase (ALT or AST) levels ≥2 times the upper limit of normal (ULN) during screening;
11. Creatinine clearance (Ccr) <45 mL/min (based on the Cockcroft-Gault formula) during screening;
12. Evidence of hematopoietic dysfunction during screening:

    1. Hemoglobin level <9.0 g/dL or hematocrit <30%;
    2. White blood cell count <3.0×10⁹/L or absolute neutrophil count (ANC) <1.2×10⁹/L;
    3. Platelet count <100×10⁹/L;
13. Abnormal 12-lead ECG findings at screening or baseline that, in the investigator's judgment, may increase the safety risk of the study intervention or affect the interpretation of study results;
14. Uncontrolled hypertension with systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥90 mmHg at screening/baseline;
15. Body mass index (BMI) >30 kg/m² during screening;
16. Contraindications to MRI, including but not limited to the presence of cardiac pacemakers, stents, artificial heart valves, etc.;
17. Subjects with a current psychiatric disorder such as anxiety or depression, or a history of such disorders, and who are deemed by the investigator to be unsuitable for participation in the study;
18. Subjects with a history of malignancy (except for adequately treated or excised non-metastatic basal cell or squamous cell carcinoma of the skin);
19. Pregnant or breastfeeding women, women planning to become pregnant during the study, and men planning to donate sperm during the study;
20. Use of high-dose corticosteroids (i.e., intravenous or intramuscular corticosteroids or oral prednisone equivalent >10 mg/day) or unstable doses (regardless of treatment for rheumatoid arthritis or other conditions) within 28 days prior to the baseline visit;
21. Subjects with a history of hypersensitivity to any component of the study intervention or similar compounds;
22. Participation in another interventional clinical study within 4 weeks prior to the baseline visit or within 5 half-lives of the last dose of the investigational drug at baseline;
23. History of alcohol or drug abuse within 6 months prior to the start of study intervention treatment, deemed by the investigator to hinder study participation;
24. Receipt of any live virus vaccination within 8 weeks prior to the baseline visit;
25. Subjects classified as legally disabled according to the April 2008 version of the "Law of the People's Republic of China on the Protection of Persons with Disabilities";
26. Subjects with potential health, mental, or social conditions that, in the investigator's judgment, may prevent or hinder compliance with the study protocol;
27. Peripheral or central nervous system disorders that, in the investigator's judgment, may interfere with the assessment of knee pain and function, such as fibromyalgia, significant low back pain, hip pain, sciatica, lumbar disc herniation, etc.;
28. Any other condition that is deemed by the investigator to be unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
TEAEs and SAEs | Within 24 weeks after the injection of hiSCs
  The incidence of TEAEs and SAEs related to the study intervention
WOMAC | At 24 weeks after the injection of hiSCs
  The change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score (range: 0-240 cm; including pain, stiffness, and physical function subscales) for the target knee, as assessed by the subject, with higher scores indicating greater symptom severity and worse physical function
GSUS | At 24 weeks after the injection of hiSCs
  The change from baseline in Gray-scale ultrasound (GSUS) (range: 0-12; including suprapatellar, medial, lateral, and posterior planes) for the target knee, as assessed by musculoskeletal ultrasound, with higher scores indicating more severe synovitis
PDUS | At 24 weeks after the injection of hiSCs
  The change from baseline in Power Doppler Ultrasound Synovitis (PDUS) score (range: 0-15; including suprapatellar, infrapatellar, medial, lateral, and posterior compartments) for the target knee, as assessed by power Doppler ultrasound, with higher scores indicating more severe synovitis

SECONDARY OUTCOMES:
ACR20, ACR50, ACR70 | At Weeks 2, 4, 8, 12, and 24
  The proportion of subjects who achieved ACR20, ACR50, and ACR70(American College of Rheumatology 20%/50%/70% improvement)
TJC | At Weeks 2, 4, 8, 12, and 24
  Change from baseline in 68-joint tender joint count (TJC; American College of Rheumatology [ACR] Core Set measure; range 0-68, higher scores indicate worse disease activity)
SJC | At Weeks 2, 4, 8, 12, and 24
  Change from baseline in 66-joint swollen joint count (SJC; ACR Core Set measure; range 0-66, higher scores indicate worse disease activity)
HAQ-DI | At Weeks 2, 4, 8, 12, and 24
  Change from baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI; ACR Core Set measure; range 0-3, higher scores indicate worse functional status)
Patient-reported pain intensity (VAS） | At Weeks 2, 4, 8, 12, and 24
  Change from baseline in patient-reported pain intensity (Visual Analog Scale [VAS]; ACR Core Set measure; 0-100 mm, higher scores indicate severe pain)
Patient-reported global disease activity (VAS) | At Weeks 2, 4, 8, 12, and 24
  Change from baseline in patient-reported global disease activity (VAS; ACR Core Set measure; 0-100 mm, higher scores indicate worse status)
Physician-evaluated global disease activity (VAS) | At Weeks 2, 4, 8, 12, and 24
  Change from baseline in physician-evaluated global disease activity (VAS; ACR Core Set measure; 0-100 mm, higher scores indicate worse status)
Acute-phase reactant | At Weeks 2, 4, 8, 12, and 24
  Change from baseline in acute-phase reactant (C-reactive protein [CRP; high-sensitivity assay; 0-10 mg/L] or erythrocyte sedimentation rate [ESR; 0-15 mm/h]; ACR Core Set measure; higher values indicate worse inflammation)
DAS28 (CRP or ESR) score of <2.6 and <3.2 | At Weeks 2, 4, 8, 12, and 24
  The proportion of subjects achieving a DAS28 (CRP or ESR) score of <2.6 and <3.2
DAS28 (CRP or ESR) | At Weeks 2, 4, 8, 12, and 24
  The change from baseline in Disease Activity Score 28 (DAS28) using C-reactive protein (CRP) or erythrocyte sedimentation rate (ESR), with higher scores indicating greater disease activity
SDAI score of ≤3.3 | At Weeks 2, 4, 8, 12, and 24
  The proportion of subjects achieving Simplified Disease Activity Index (SDAI) remission (score ≤3.3; total score range: 0-86), with lower scores indicating better disease control
SDAI | At Weeks 2, 4, 8, 12, and 24
  The change from baseline in Simplified Disease Activity Index (SDAI)score（total score range: 0-86), with lower scores indicating better disease control
CDAI score of ≤2.8 | At Weeks 2, 4, 8, 12, and 24
  The proportion of subjects achieving Clinical Disease Activity Index (CDAI) remission (score ≤ 2.8; total score range: 0-76), with lower scores indicating better disease control
CDAI | At Weeks 2, 4, 8, 12, and 24
  The change from baseline in Clinical Disease Activity Index (CDAI)score (total score range: 0-76), with lower scores indicating better disease control
VAS | At Weeks 2, 4, 8, and 12
  The change from baseline in Visual Analog Scale (VAS) score (range: 0-100 mm) for the target knee, as assessed by the subject, with higher scores indicating greater symptom severity and worse physical function
WOMAC | At Weeks 2, 4, 8, and 12
  The change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score (range: 0-240 cm; including pain, stiffness, and physical function subscales) for the target knee, as assessed by the subject, with higher scores indicating greater symptom severity and worse physical function
KOOS | At Weeks 2, 4, 8, 12, and 24
  The change from baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS) (range: 0-100; including Pain, Symptoms, Activities of Daily Living, Sport/Recreation, and Quality of Life subscales), as assessed by the subject, with higher scores indicating better function and fewer symptoms
WORMS | At 24 weeks after the injection of hiSCs
  The change from baseline in Whole-Organ Magnetic Resonance Imaging Score (WORMS) (assessing ：cartilage morphology [0-6 per subregion], bone marrow lesions [0-3 per subregion], meniscal pathology [0-4 per meniscus], subchondral cysts [0-3 per subregion], osteophytes [0-7 per subregion], bone attrition [0-3 per subregion], synovitis [0-3], ligament abnormalities [0-2 per ligament], periarticular cysts [0-3], and loose bodies [0-3]), as assessed by MRI, with higher scores indicating more severe structural damage
MOAKS | At 24 weeks after the injection of hiSCs
  The change from baseline in the MRI Osteoarthritis Knee Score (MOAKS) (assessing: cartilage damage [0-3 per subregion], bone marrow lesions [0-3 per subregion], osteophytes [0-3 per subregion], meniscal pathology [0-5 per meniscus], synovitis/effusion [0-3], ligament/tendon abnormalities [0-1 per ligament/tendon], and periarticular features [0-1]), as assessed by MRI, with higher scores indicating more severe structural damage
BLOKS | At 24 weeks after the injection of hiSCs
  The change from baseline in the Boston-Leeds Osteoarthritis Knee Score (BLOKS) (assessing: cartilage morphology [0-3 per region, cartilage area loss；0-2 per region, thickness loss], bone marrow lesions [0-3 per region], osteophytes [0-3 per region], meniscal pathology [0-5 per meniscus], synovitis/effusion [0-3], ligament abnormalities [0-1 per ligament], and periarticular features [0-1]), as assessed by MRI, with higher scores indicating more severe structural damage
Synovial thickness | At 24 weeks after the injection of hiSCs
  The change from baseline in synovial thickness (mm), as assessed by MRI, with increased values indicating greater synovial inflammation
Synovial blood flow | At 24 weeks after the injection of hiSCs
  The change from baseline in synovial blood flow (measured in mL/min/100g tissue), as assessed by MRI, with increased values indicating greater vascularity
Joint effusion volume | At 24 weeks after the injection of hiSCs
  The change from baseline in joint effusion volume(mL), as assessed by MRI, with increased values indicating greater effusion severity
GSUS | At Weeks 2, 4, 8, and 12
  The change from baseline in Gray-scale ultrasound (GSUS) (range: 0-12; including suprapatellar, medial, lateral, and posterior planes) for the target knee, as assessed by musculoskeletal ultrasound, with higher scores indicating more severe synovitis
PDUS | At Weeks 2, 4, 8, and 12
  The change from baseline in Power Doppler Ultrasound Synovitis (PDUS) score (range: 0-15; including suprapatellar, infrapatellar, medial, lateral, and posterior compartments) for the target knee, as assessed by power Doppler ultrasound, with higher scores indicating more severe synovitis

OTHER OUTCOMES:
Cytomorphology | At 4 weeks after the injection of hiSCs
  The change from baseline in synovial fluid morphological characteristics (%) in the target knee, as assessed by pathological microscopy
Total protein | At 4 weeks after the injection of hiSCs
  The change from baseline in synovial fluidtotal protein concentration (g/L) in the target knee
Cytokine response | At 4 weeks after the injection of hiSCs
  The change from baseline in synovial fluid cytokine response（large panel of cytokines characteristic of the inflammatory response, including TNFα, IL-6, IL-8, IL-10, γ-IFN, IL-17A, SERPINA3, TGFβ1, IGFBP7, MMP-3, VEGF) in the target knee
RF | At 4 weeks after the injection of hiSCs
  The change from baseline in synovial fluidrheumatoid factor (RF) concentration (IU/ML) in the target knee

CONTACTS AND LOCATIONS:
Overall Officials: Huji Xu, Ph.D, MD, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai ChangZheng hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Due to concerns about the security of patients' personal information